CLINICAL TRIAL: NCT03103828
Title: Promoting Healthcare Planning as a Healthy Behavior (STAMP VA)
Brief Title: Sharing and Talking About my Preferences
Acronym: STAMPVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TF0025
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Computer-tailored intervention (Active Comparator)
  Interventions: Behavioral: Computer-Tailored Intervention
- Motivational Interviewing (Active Comparator)
  Interventions: Behavioral: Motivational Interviewing
- Motivational Enhancement Therapy (Active Comparator)
  Interventions: Behavioral: Motivational Enhancement Therapy
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Computer-Tailored Intervention — CTI will receive telephone contact at three time points: baseline, two, and four months. Each contact consists of an integrated assessment and intervention feedback report, using an expert system. Participants are assessed for four different behaviors that together represent complete ACP engagement: communication with loved ones about views on quality of life versus quantity of life, communication with clinicians about views on quality of life versus quantity of life, assignment of a health care surrogate, and completion of a living will. The system takes the results of the assessment and results in an individualized feedback report.
  Arms: Computer-tailored intervention
Behavioral: Motivational Interviewing — MET will receive telephone contact at three time points: baseline, two, and four months. They will undergo the assessment as described above receive and they will receive a second a telephone contact within two weeks of the assessment, which will consist of an MET session. If the surrogate has been enrolled in the study, the MET will be conducted with both the Veteran and the surrogate in a dyadic telephone interview. The goal of the interview is to strengthen commitment to engage in ACP and promote self-efficacy. The interviewer will also help the Veteran to reflect on the pros and cons of ACP engagement as elicited in the assessment process, to understand how to build on ACP behaviors already engaged in, and, if appropriate, to help the Veteran create a change plan for further ACP engagement.
  Arms: Motivational Interviewing
Behavioral: Motivational Enhancement Therapy — Participants assigned to CTI+MET will receive the CTI intervention at baseline, two months, and four months as described above. with a follow-up MET session as described above occurring within two weeks of each contact.
  Arms: Motivational Enhancement Therapy

SUMMARY:
The purpose of this study is to figure out the best way to help veterans do advance care planning. This study will examine the effects of two theory based behavior interventions by randomizing veteran into 4 groups to see which veterans will complete the 4 step process of advance care planning.

DETAILED DESCRIPTION:
Purpose: The purpose of this study is to examine the effects of two theory-based behavior interventions on engagement of Veterans in advance care planning (ACP) by means of the following specific aim:

Primary Aim: To conduct a randomized controlled trial examining the effects of: a) usual care; b) computer-tailored intervention (CTI); c) motivational enhancement therapy (MET); d) CTI + MET on the proportion of middle-age and older Veterans receiving primary care at the VA who complete the process of ACP, defined as completing a total of 4 key ACP behaviors, including selecting a health care proxy, communicating with the proxy about goals of care, communicating with the clinician about goals of care, and documenting proxy selection and goals.

Primary Hypothesis: The proportion of Veterans completing ACP will be higher among those in each of the intervention groups compared to Veterans receiving usual care.

All of 4 groups will receive their assessments and, if, their interventions, by telephone and/or mail. The veterans will from the VA Connecticut Healthcare System. Participants will be identified through a data query of the Regional Data Warehouse who have had a primary care visit in the past 12 months. We will then be able to oversample female and minority Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Veteran

  ---Must have seen primary care provider in the past 12 months
* Primary language is English

Exclusion Criteria:

* Severe hearing or vision loss

  * moderate-to-severe cognitive impairment
* active psychiatric illness
* No regular phone or permanent address

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 484 (Estimated)
Dates: Start 2017-10-02 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Completion of 4 ACP behaviors | 6 months
  Having completed 4 ACP behaviors: living will, health care agent, communication with loved ones about quality versus quantity of life, having forms in medical record

SECONDARY OUTCOMES:
Movement on each of 4 ACP behaviors | 6 months
  Progression in readiness to change for each of the 4 ACP behaviors described above.

CONTACTS AND LOCATIONS:
Overall Officials: Terri Fried, MD, Principal Investigator — VAConnecticut Healthcare System
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fried TR, Yang M, Martino S, Iannone L, Zenoni M, Blakley L, O'Leary JR, Redding CA, Paiva AL. Effect of Computer-Tailored Print Feedback, Motivational Interviewing, and Motivational Enhancement Therapy on Engagement in Advance Care Planning: A Randomized Clinical Trial. JAMA Intern Med. 2022 Dec 1;182(12):1298-1305. doi: 10.1001/jamainternmed.2022.5074. PMID 36342678
- [Derived] Fried TR, Redding CA, Martino S, Paiva A, Iannone L, Zenoni M, Blakley LA, Rossi JS, O'Leary J. Increasing engagement in advance care planning using a behaviour change model: study protocol for the STAMP randomised controlled trials. BMJ Open. 2018 Aug 10;8(8):e025340. doi: 10.1136/bmjopen-2018-025340. PMID 30099405